CLINICAL TRIAL: NCT07308431
Title: The Effect of Single-leg 20-degree Squats Combined With Conventional Training on the Biomechanical Characteristics of Gait After Anterior Cruciate Ligament Reconstruction Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20250156
Record Dates: First submitted 2025-09-01; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Both groups underwent conventional training. In addition, the experimental group underwent single-leg 20° squat training. Participants were required to stand for the exercise and hold onto a stable surface with their hands, while the unaffected lower limb hip joint was extended and the knee joint flexed to 90°. Participants were then instructed to bend the affected knee to 20° and hold this position for 10 seconds. They then fully extended the knee and rested in that position for 3-4 seconds. The load form can be dumbbells.
  Interventions: Behavioral: single-leg 20° squat training
- control group (Active Comparator): In the 1-8 week rehabilitation program, the goal is to strengthen the muscle strength of the affected knee joint and gradually introduce functional movement exercises, while avoiding forceful flexion and extension of the knee. The specific rehabilitation program includes: prone leg curl exercises, quadriceps resistance band training, hamstring progressive resistance exercises, backward lunge exercises, in-place small jumps, knee joint flexion with appropriate cushioning, in-place squat jumps, landing and immediately squatting for stability, repeated 15 times, each lasting 2-3 seconds, performed 2-3 sets per week, totaling 3 sessions; Wall-supported static squat exercises, repeated 5 times, performed 2-3 sets per week, totaling 3 sessions.
  Interventions: Behavioral: regular training

INTERVENTIONS:
Behavioral: single-leg 20° squat training — Both groups underwent conventional training. In addition, the experimental group underwent single-leg 20° squat training. Participants were required to stand for the exercise and hold onto a stable surface with their hands, while the unaffected lower limb hip joint was extended and the knee joint flexed to 90°. Participants were then instructed to bend the affected knee to 20° and hold this position for 10 seconds. They then fully extended the knee and rested in that position for 3-4 seconds. The load form can be dumbbells.
  Arms: experimental group
Behavioral: regular training — In the 1-8 week rehabilitation program, the goal is to strengthen the muscle strength of the affected knee joint and gradually introduce functional movement exercises, while avoiding forceful flexion and extension of the knee. The specific rehabilitation program includes: prone leg curl exercises, quadriceps resistance band training, hamstring progressive resistance exercises, backward lunge exercises, in-place small jumps, knee joint flexion with appropriate cushioning, in-place squat jumps, landing and immediately squatting for stability, repeated 15 times, each lasting 2-3 seconds, performed 2-3 sets per week, totaling 3 sessions; Wall-supported static squat exercises, repeated 5 times, performed 2-3 sets per week, totaling 3 sessions.
  Arms: control group

SUMMARY:
Anterior cruciate ligament (ACL) tears are one of the most common sports injuries, with an ACL injury rate as high as 20.9% in the general population . Currently, the primary treatment for ACL tears is arthroscopic reconstruction surgery to restore knee stability and function . Following ACL injury, abnormal gait biomechanical characteristics persist, even after ACL reconstruction surgery (ACLR) and evidence-based rehabilitation therapy. These abnormal gait biomechanical characteristics remain unresolved, with the lower limbs exhibiting insufficient loading and stiffness, which are associated with quadriceps muscle dysfunction. Interventions for quadriceps atrophy following ACLR should be initiated early to prevent worsening of early knee pain, swelling, and abnormal gait. Additionally, since ACL reconstruction results in different biomechanical characteristics at various stages and gait phases, it is important to adopt more targeted and precise rehabilitation measures to correct biomechanical abnormalities and improve gait function in patients.

DETAILED DESCRIPTION:
Research Background: The anterior cruciate ligament (ACL) is one of the important anatomical structures in the knee joint, maintaining knee stability and preventing anterior displacement of the tibia. Following ACL injury, abnormal gait biomechanical characteristics persist, even after ACL reconstruction surgery (ACLR) and evidence-based rehabilitation therapy, with abnormal gait biomechanics failing to fully recover. Quadriceps atrophy is a common cause of abnormal gait biomechanics and persists long-term postoperatively. The quadriceps are closely related to knee joint function and contribute most significantly to knee joint stability and movement control. Therefore, intervention for quadriceps atrophy following ACLR should be initiated early to prevent worsening of early knee pain, swelling, and abnormal gait. Post-ACLR rehabilitation aims to protect the graft, promote its biological remodeling, and limit the extent of muscle atrophy while facilitating muscle strength recovery. Additionally, since ACL injury and reconstruction exhibit different biomechanical characteristics at various stages and gait phases, it is essential to adopt more targeted and precise rehabilitation measures to correct biomechanical abnormalities and improve gait function. Research methods: This study plans to recruit 48 patients 12 weeks post-ACL reconstruction surgery, divided into an experimental group and a control group. The experimental group will undergo single-leg mini squat (SLMS) training in addition to conventional training, with kinematic and dynamic data collected simultaneously using a three-dimensional motion capture system and force plate system; electromyographic signals will be collected from patients during gait testing. Additionally, three-dimensional finite element modeling will be used to calculate the stress distribution and peak stress on the ACL graft during SLMS. Expected Study Outcomes: This study anticipates that after 8 weeks of SLMS training, the knee flexion angle during the stance phase of walking, knee extension torque, and activity of the medial femoral muscle during walking will increase. Additionally, the study aims to confirm that SLMS training keeps stress on the ACL graft within a safe range.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unilateral Anterior Cruciate Ligament (ACL) rupture.
* Aged between 18 and 45 years.
* Scheduled for primary unilateral ACL reconstruction at our hospital.
* Presence of quadriceps atrophy, defined as the bilateral difference in quadriceps strength is >10% of the contralateral unaffected limb.
* The operated knee has no significant redness, swelling, pain, inflammation, or limitations in range of motion and has essentially restored basic joint mobility.
* No or only minor (Grade I) injury to the posterior cruciate ligament, medial collateral ligament, or lateral collateral ligament.

Exclusion Criteria:

* Severe injury (Grade II or III) to the posterior cruciate ligament, medial collateral ligament, or lateral collateral ligament in the affected knee.
* Concomitant severe meniscal tear(s) in the affected knee.
* History of significant prior trauma or surgery to the affected knee.
* Presence of other knee joint diseases (e.g., osteoarthritis, tumors, rheumatoid arthritis, tuberculosis).
* Poor subject compliance or anticipated inability to complete the entire study protocol.Subject withdrawal of informed consent.
* Any reason the subject proposes to terminate the study or is unable to complete the trial.
* In the investigator's judgment, continued participation would adversely affect the subject's physical condition.
* Decision by the Ethics Review Committee to terminate the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Knee joint kinematics during walking | Assessed at 12 weeks post-operation and again after 8 weeks of intervention (total assessment period of 2 months）
  Kinematic angles (flexion, rotation, and adduction) of the knee joint in the sagittal, frontal, and horizontal planes during walking.
Knee joint kinetics during walking | Assessed at 12 weeks post-operation and again after 8 weeks of intervention (total assessment period of 2 months)]
  The moment generated at the knee joint during walking.
Gait-Synchronized Electromyographic Signals | Assessed at 12 weeks post-operation and again after 8 weeks of intervention (total assessment period of 2 months)]
  Outcome Measure 1: Raw electromyographic (EMG) activity Raw EMG signals of the rectus femoris, vastus lateralis, vastus medialis, biceps femoris, and semitendinosus muscles during specified movements.
  Outcome Measure 2: Integrated electromyographic (IEMG) activity The integrated EMG (IEMG) of the rectus femoris, vastus lateralis, vastus medialis, biceps femoris, and semitendinosus muscles during specified movements.
  Outcome Measure 3: Average electromyographic (AEMG) amplitude The average EMG amplitude (AEMG) of the rectus femoris, vastus lateralis, vastus medialis, biceps femoris, and semitendinosus muscles during specified movements.
Isokinetic muscle strength | Assessed at 12 weeks post-operation and again after 8 weeks of intervention (total assessment period of 2 months)
  Quadriceps isokinetic strength test: Isokinetic biomechanical test and trainer (CON-TREX, MJ; Germany), conducted by the same tester on a constant velocity device. Three complete movements need to be collected, with an interval of 90 seconds between each test to avoid fatigue. The quadriceps muscle was tested for isokinetic and eccentric peak torque (PT) at 60°/s.
Anterior cruciate ligament stress distribution and peak. | Completed through study, averaging 3 months.
  * Joint flexion, rotation and adduction angles of the knee joint in the sagittal, frontal and horizontal planes during walking and squatting at 20°.
  * measured during squatting at 12 weeks post-anterior cruciate ligament reconstruction surgery. Stress and strain distribution in the anterior cruciate ligament at a 20-degree squat angle were calculated using ANSYS.
Anterior cruciate ligament stress distribution and peak. | "through study completion, an average of 3 month".
  * the moment generated during movement, and the tibial displacement during squats at 20°.
  * measured during squatting at 12 weeks post-anterior cruciate ligament reconstruction surgery. Stress and strain distribution in the anterior cruciate ligament at a 20-degree squat angle were calculated using ANSYS.

SECONDARY OUTCOMES:
Lysholm Knee Scoring Scale | Assessed at 12 weeks post-operation and again after 8 weeks of intervention (total assessment period of 2 months)]
  The Lysholm Knee Scoring Scale, a patient-reported outcome measure assessing knee function. Scores range from 0 to 100, where higher scores indicate a better outcome.
International Knee Documentation Committee Subjective Knee Form | Assessed at 12 weeks post-operation and again after 8 weeks of intervention (total assessment period of 2 months）
  The International Knee Documentation Committee Subjective Knee Form, a patient-reported outcome measure assessing symptoms, function, and sports activity. Scores range from 0 to 100, where higher scores indicate a better outcome.
Thigh circumference measurement | Assessed at 12 weeks post-operation and again after 8 weeks of intervention (total assessment period of 2 months)
  The circumference of the thigh, measured at a standardized anatomical location, to assess muscle atrophy or swelling. A smaller circumference indicates a worse outcome (greater atrophy or reduced swelling).

IPD SHARING:
Plan to Share IPD: No